CLINICAL TRIAL: NCT07004842
Title: Alternative Carer Respite: A Study on Its Effectiveness and Potential Mechanisms
Brief Title: Alternative Carer Respite: A Study on Its Effectiveness and Potential Mechanism
Acronym: VRDCFIn-home1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Vivian W.Q. Lou, Director, Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EA230565
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Caregiver Burden
Keywords: respite; caregiver burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregivers (Experimental): Caregivers will receive 48 hours of respite service within 6 months
  Interventions: Other: 48 hr Respite Service

INTERVENTIONS:
Other: 48 hr Respite Service — Caregivers will be provided with 48 hours of respite service within 6 months. Trained alternative caregivers will provide elderly-sitting service at their home, allowing the caregivers to have their personal time.

SUMMARY:
The primary objective of this study is to examine the effectiveness of alternative carer respite in meeting the unique needs of older adults without children or with limited contact with their children in Hong Kong. Caregivers are assessed before and after the intervention, and three months after the end of intervention on their physical health, mental well-being, social engagement, and overall satisfaction.

DETAILED DESCRIPTION:
All participants will provide informed consent at the time of enrolment. Both caregivers and their care recipients will complete an assessment. Caregivers are screened for their physical health, mental well-being, social engagement, and overall satisfaction. Care recipients are screened using InterRAI for their physical functions.

Caregivers will receive a maximal of 48 hours of respite service within 6 month. Alternative caregivers will provide in-home elderly-sitting service so that the caregivers can have some private time for themselves.

At the end of the service period, caregivers and care recipients will complete the assessment again to measure the changes of their physical and mental health.

All participants will be contacted again for follow-up assessment 3 months after the completion of service.

ELIGIBILITY:
Inclusion Criteria:

* Either the CR or CG is aged ≥60
* Reported having (a) no children; OR (b) no children in Hong Kong; OR (c) having children in Hong Kong but with limited contact (i.e., fewer than once per month in any forms)
* Voluntary participation.

Exclusion Criteria:

* Unable to communicate in neither Cantonese, English nor Mandarin

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in score in caregiving needs on the Carer Needs Screening Tool (CNST-11) after the intervention | Baseline and Immediate after intervention
  The Carer Needs Screening Tool (CNST-11) is a self-developed tool that measures different aspects of caregiving needs over the past 1 week period. It is a 11-item scale, with 8 items that determines the overall needs level and the others for four aspects of needs: physical health, mental health, social support and care needs. Possible score is from 8 to 32 with lower score indicates lower caregivers' needs.
  Change in score = Immediate after intervention - baseline
Change from baseline in score in depression symptoms on PHQ-9 after the intervention | Baseline and Immediate after intervention
  The Patient History Questionnaire (PHQ-9) is a widely used tool that consists of nine questions designed to screen and monitor the presence and severity of depression. The total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating more severe depressive symptoms. The score ranges for the PHQ-9 are as follows: 0-4: Minimal depression symptoms; 5-9: Mild depression; 10-14: Moderate depression; 15-19: Moderately severe depression; 20-27: Severe depression Change in score = Immediate after intervention - baseline
Change from baseline in score in anxiety symptoms on GAD-7 after the intervention | Baseline and Immediate after intervention
  The Generalized Anxiety Disorder 7 (GAD-7) involves 7- items assessing the severity of anxiety symptoms. The total score on the GAD-7 ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms. The score ranges for the GAD-7 are as follows: 0-4: Minimal anxiety symptoms; 5-9: Mild anxiety; 10-14: Moderate anxiety; 15-21: Severe anxiety.
  Change in score = Immediate after intervention - baseline
Change in score from baseline in quality of life measured by EQ-5D-5L after intervention | Baseline and Immediate after intervention
  The EQ-5D-5L is a standardized instrument used to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The responses are converted into a single index value representing overall health status using Hong Kong's normative value. The primary outcome measure in this study is the change in EQ-5D-5L index scores from baseline to post-intervention/follow-up assessments. 1 equals to perfect health and more negative numbers indicates worse health. Change in health index = Immediate after intervention - baseline
Changes in score from baseline in perception of caregiving measured by Positive Aspect of Caregiving scale after intervention | Baseline and Immediate after intervention
  The Positive Aspect of Caregiving scale is a 11-item scale that measures how the caregiver perceive caregiving experience, specifically in a positive aspect (e.g., caregiving makes me feel useful). It is rated in a 5-point Likert scale from "very disagree" to "very agree", with potential score from 0 to 44. A higher score indicates caregiving perceiving it in a more positive way.

OTHER OUTCOMES:
Retention of changes of Primary outcome 1 to 5 after the end of intervention | Baseline, immediate after intervention, 3 months after the intervention
  Caregivers will complete the primary outcome measurements (1 to 5) again 3, 6 and 12 months after the end of the intervention. They will not receive any in-home respite service from the project in between the measurement periods. Changes in score of each scale in Primary Outcome 1 to 5 will be measured. Participants with improved/sustained score indicates better retention.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Weiqun Lou, PhD, Principal Investigator — Sau Po Centre on Ageing, University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
IPD (including protocol and anonymized dataset) will be made available upon request, subject to ethical review and data protection regulations